CLINICAL TRIAL: NCT07314190
Title: Synapsing Retrospective Biomarker Study
Brief Title: Retrospective Observational Study of Blood-based Biomarkers in the Diagnosis and Monitorign of Patients With a Neurodegenerative Disease or Mental Disorder
Acronym: Synapsing-BK
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: University of Ulm (Other); University Of Perugia (Other); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Olivia E Belbin, PhD, Dr, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-ENT-2024-175; 101156566 (Other Grant/Funding Number: EU Horizon Europe)
Record Dates: First submitted 2025-11-14; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Dementia With Lewy Bodies (DLB); Frontotemporal Dementia (FTD); Major Depressive Disorder (MDD); Bipolar 1 Disorder; Schizophenia Disorder; Parkinson Disease
Keywords: Companion diagnostic biomarker; Synapse biomarker; magnetic resonance imaging; plasma; blood; serum
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia; Depressive Disorder, Major; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood (plasma and serum)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Major depressive disorder: Clinical diagnosis of major depressive disorder
- Bipolar disorder: Clinical diagnosis of type I + II Bipolar disorder
- Schizophrenia: Clinical diagnosis of schizophrenia
- Parkinson's disease: Clinical diagnosis of Parkinson's disease
- Alzheimer's disease: Clinical diagnosis of Alzheimer's disease
- Dementia with Lewy bodies: Clinical diagnosis of dementia with Lewy bodies
- Unaffected controls: No clinical diagnosis of a primary psychiatric disorder or neurodegenerative disease
- Frontotemporal dementia: Clinical diagnosis of frontotemporal dementia

SUMMARY:
This is a retrospective observational study to evaluate the clinical utility of blood-based biomarkers in the diagnosis and management of patients with a neurodegenerative disease (ND) or mental disorder (MD).

DETAILED DESCRIPTION:
This study will collect clinical and biomarker data from patients and controls to identify a) a blood-based diagnostic biomarker for mental disorders, and b) a blood-based biomarker that could be used as a surrogate end-point for the principal neuropsychiatric symptoms.

Specific research questions are:

Can blood-based biomarkers provide a faster more objective diagnosis for major depressive disorder, bipolar disorders or schizophrenia? Can the same biomarkers also aid in the differential diagnosis from neurodegenerative diseases? Do blood-based synaptic biomarkers correlate with structural and functional brain changes, cognitive performance and psychiatric symptoms in patients with major depressive disorder, bipolar disorders, schizophrenia, Alzheimer's disease, dementia with Lewy bodies, frontotemporal dementia or Parkinson's disease? Can the blood-based synaptic biomarkers predict therapeutic response in patients with major depressive disorder, bipolar disorders or schizophrenia?

ELIGIBILITY:
Inclusion Criteria:

* Age>18 and donation of blood,
* full clinical and psychological assessment
* Available neuroimaging is optional as not all patients are suitable.
* Age and sex-matched unaffected volunteers without a MD or ND diagnosis are used as controls.
* Unaffected controls are usually spouses or children of patients that are informed about our studies at each clinical site.

Exclusion Criteria:

* Lack of neuropsychological data,
* anticoagulant treatment such as acenocoumarol, heparin, warfarin, dabigatran, rivaroxaban, apixaban, drug abuse in the last year,
* medical history of cancer affecting the central nervous system that has not been in complete remission for 5 years or longer,
* the patient has received potentially neurotoxic chemotherapy and/or patient has received cranial radiotherapy.
* Clinical diagnosis of Alzheimer's disease where pathophysiological markers (measured in CSF or plasma) are inconsistent with Alzheimer's disease pathophysiology.
* Cognitively healthy volunteers where pathophysiological markers (measured in CSF or plasma) are consistent with Alzheimer's disease or other neurodegenerative pathophysiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from specialized clinics at Barcelona (Spain), Perugia (Italy), Ulm (Germany), Halle (Germany) and Kuopio (Finland). Target % female in schizophrenia (30%), major depressive disorder (50%), bipolar disorder and controls (55%), Alzheimer's disease and controls (60%), frontotemporal dementia (65%), controls (65%). These percentages match those typically found in these disorders. Unaffected controls are usually spouses or children of patients that are informed about our studies at each clinical site.
Sampling Method: Non-Probability Sample
Enrollment: 1799 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of biomarkers in blood | through study completion, an average of 1 year
  Concentration of biomarker (eg., NPTX2) in blood measured by immunoassay or mass spectrometry-based techniques.
Diagnosis | Baseline
  Primary diagnosis following evaluation by clinician and neuropsychologist
Boston Naming Test | Up to 3-months
  Total score on the Boston Naming Test

SECONDARY OUTCOMES:
Structural brain changes | Up to 3-months
  Acquisition of 3T-MRI with a high-resolution 3D T1-weighted anatomical image, a multi-shell diffusion-weighted MRI, and a resting-state functional sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau - IIB Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No